CLINICAL TRIAL: NCT05174390
Title: Thumb ECG IncidenT Atrial fibrillatioN in Diabetes Mellitus
Acronym: TITAN-DM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Gävleborg (Other)
Responsible Party: Sponsor
Other Study IDs: 202103323
Record Dates: First submitted 2021-11-30; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus; Atrial Fibrillation
Keywords: atrial fibrillation; diabetes mellitus; thumb-ECG
MeSH Terms: conditions — Diabetes Mellitus; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coala Heart Monitor Pro — thumb- and chest-ECG

SUMMARY:
Cardiac thromboembolism attributed to atrial fibrillation (AF) constitutes at least one-third of ischemic strokes. Indeed, stroke may be the first manifestation of previously undetected AF. The prevalence is projected to increase 20% the coming decades, especially in age group 65 years and above of age. To add to incidence, the diabetic population have an increased risk yet not properly investigated. In patients with confirmed AF, assessment using the CHA2DS2-VASc score (congestive heart failure, hypertension, age 65 years and above, diabetes mellitus, stroke, vascular disease, age 75 years and above, sexual category), is applied for risk stratification. If the CHA2DS2-VASc score is at least 1, or definitely 2 points typically a non-vitamin K antagonist oral anticoagulant (NOAC) should be prescribed. The chest- and thumb-electrocardiogram (ECG) system Coala Heart Monitor has proven efficacious in detecting AF following recent cryptogenic stroke. This system also showed to be feasible from a patient perspective. Thus, in patients aged 65 years and above with diabetes mellitus at least 2 points are reached. Therefore, patient with these risk factors should be considered for further evaluation for NOAC to prevent stroke, which provides the rational for this study.

DETAILED DESCRIPTION:
Cardiac thromboembolism attributed to atrial fibrillation (AF) constitutes at least one-third of ischemic strokes.The prevalence is projected to increase 20% the coming decades, especially in age group 65 years and above of age. To add to incidence, the diabetic population have an increased risk yet not properly investigated. In patients with confirmed AF, assessment using the CHA2DS2-VASc score (congestive heart failure, hypertension, age 65 years and above, diabetes mellitus, stroke, vascular disease, age 75 years and above, sexual category) , is applied for risk stratification. If the CHA2DS2-VASc score is at least 1, or definitely 2 points typically a Non-vitamin K antagonist Oral AntiCoagulants (NOAC) should be prescribed. The chest- and thumb-electrocardiogram (ECG) system Coala Heart Monitor will be used to detect AF, which showed to be feasible from a patient perspective. Thus, in patients aged 65 years and above with diabetes mellitus at least 2 points are reached. Therefore, patient with these risk factors should be considered for further evaluation for NOAC to prevent stroke, which provides the rational for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and above
* Diabetes mellitus (both type 1 and type 2)

Exclusion Criteria:

* Treatment with anticoagulation (Eliquis, Lixiana, Pradaxa, Xarelto, Waran)
* Pacemaker, implantable cardioverter defibrillator, insertable cardiac monitor
* Not able to participate in 90 days follow-up

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Unselected patients with diabetes type 1 or type 2 at an age of 65 years and above.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the diagnosis of atrial fibrillation | 90 days
  Incidence of atrial fibrillation during the monitoring period

SECONDARY OUTCOMES:
Patient-reported symptoms (descriptive category variables) of atrial fibrillation using a questionnaire in a digital application | 90 days
  Symptoms (questionnaire with the following categories of answers: palpitation, dizziness, dyspnea, chest pain, other) when atrial fibrillation is diagnosed using the patient report (in the digital application with the mentioned categories of symptoms predefined) at the time of ECG transmission.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Gavleborg, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Magnusson P, Lyren A, Mattsson G. Patient-reported feasibility of chest and thumb ECG after cryptogenic stroke in Sweden: an observational study. BMJ Open. 2020 Oct 28;10(10):e037360. doi: 10.1136/bmjopen-2020-037360. PMID 33115891